CLINICAL TRIAL: NCT00499122
Title: Phase II Study of Neoadjuvant Treatment With NOV-002 in Combination With Doxorubicin and Cyclophosphamide Followed by Docetaxel in Patients With Stages IIB-IIIC Breast Cancer
Brief Title: NOV-002, Doxorubicin, Cyclophosphamide, and Docetaxel in Women With Newly Diagnosed Stage II or IIIC Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20071167; MUSC-101072 (Other: Medical University of South Carolina); MUSC-HR-17111 (Other: Medical University of South Carolina)
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2013-03-29 (Estimated); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Breast Cancer
Keywords: stage II breast cancer; stage IIIC breast cancer; inflammatory breast cancer
MeSH Terms: conditions — Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Cyclophosphamide; Docetaxel; Doxorubicin; NOV 002; Glutathione Disulfide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NOV-002 and Chemotherapy (Experimental): * NOV-002:
    * Cycle 1, Day -1 only: 60 mg intravenously (IV) x 2, 3 hours (+/- 30 minutes) apart
    * Cycles 1 - 8, Day 1: 60 mg IV, 1 hour (+/- 30 minutes) prior to chemotherapy administration
    * Cycle 1 - 8, Days 2 - 21: 60 mg subcutaneous injections
  * Cyclophosphamide: 600 mg/m2 IV, Cycles 1 - 4, Day 1
  * Doxorubicin: 60 mg/m2 IV, Cycles 1 - 4, Day 1
  * Docetaxel: 100 mg/m2 IV, Cycles 5 - 8, Day 1
  Interventions: Drug: Cyclophosphamide; Drug: Docetaxel; Drug: Doxorubicin; Drug: NOV 002

INTERVENTIONS:
Drug: Cyclophosphamide
  Other Names: Cytoxan
Drug: Docetaxel
  Other Names: Cytoxan
Drug: Doxorubicin
  Other Names: Adriamycin
Drug: NOV 002
  Other Names: Oxidized glutathione

SUMMARY:
RATIONALE: Oxidized glutathione (NOV-002) may stimulate the immune system in different ways and stop tumor cells from growing. Drugs used in chemotherapy, such as doxorubicin, cyclophosphamide, and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells. Giving NOV-002 together with chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

PURPOSE: This phase II trial is studying how well giving oxidized glutathione (NOV-002) together with doxorubicin and cyclophosphamide followed by docetaxel works in treating women with newly diagnosed stage II or stage III breast cancer.

DETAILED DESCRIPTION:
OUTLINE: This is a multicenter study.

Patients receive oxidized glutathione (NOV-002) IV twice on day -1 of course 1 and once on day 1 of courses 2-8. Patients receive NOV-002 subcutaneously once daily on days 2-21 of courses 1-8. Patients also receive chemotherapy comprising doxorubicin hydrochloride IV and cyclophosphamide IV on day 1 of courses 1-4 followed by docetaxel IV on day 1 of courses 5-8. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients undergo definitive surgery 3-6 weeks after completion of neoadjuvant therapy.

Blood samples are obtained at baseline and periodically during study to measure serum and plasma protein glutathionlylation. Additional blood samples are collected from some patients for immunological correlative studies.

After completion of study therapy, patients are followed at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Females age 18 years or older.
* The ability to provide written informed consent prior to study specific screening procedures, with the understanding that the patient has the right to withdraw from the study at any time.
* Histologically confirmed infiltrating (invasive) breast cancer by core needle biopsy, with no evidence of metastatic disease except to the ipsilateral axillary lymph nodes.
* Clinical stage IIB - IIIC (T2-4, N0 or N1, M0 or - any T, N1-3, M0) breast cancer. The primary tumor must be greater than or equal to 2 cm (T2-4) or with pathologically proven axillary nodal involvement (N1-3).
* Patients with inflammatory breast cancer (T4) are permitted into the study.
* Clinically palpable tumor that meets the criteria of RECIST for palpable measurable disease. The primary tumor must be greater than or equal to 2 cm (T2-4) or with pathologically proven axillary nodal involvement (N1-3). Bilateral synchronic breast cancers are allowed but one of the primary tumors should be selected as the target tumor.
* Primary tumor may be estrogen or progesterone receptor negative or positive, and human epidermal growth factor receptor 2 (HER-2/neu) negative as determined by either Fluorescent In Situ Hybridization (FISH) or 0-2+ staining by immunohistochemistry (IHC) (Hercept™).
* Normal cardiac ejection fraction (EF ≥ 50%) as determined by screening multigated acquisition scan (MUGA) or echocardiogram.
* No prior history of myocardial infarction, congestive heart failure, symptomatic coronary artery disease, or cardiac arrhythmias.
* Patients must be ambulatory with Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* The patient or her caregiver must be able to self administer daily subcutaneous injections.
* Life expectancy greater than 6 months.

Exclusion Criteria:

* Prior therapy of any modality for the treatment of breast cancer
* Any prior therapy with an anthracycline or a taxane for any other indication
* HER-2 positive breast cancer defined as either gene amplification by Fluorescent In Situ Hybridization (FISH) or 3+ staining by IHC (Hercept™).
* Women who have a positive pregnancy test, no pregnancy test available, who are pregnant or who are lactating.
* Women of childbearing potential must agree to use a reliable and appropriate contraceptive method, which could include a double barrier method (condom plus diaphragm), an intrauterine device or oral contraceptives. Women with ER or PR positive breast cancer, should not, however, use oral contraceptives as a method of contraception. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Women with breast cancer that do not have palpable breast tumors at screening.
* History of another malignancy within the last 5 years except curatively treated basal cell carcinoma of the skin or cervical intraepithelial neoplasia.
* Clinically significant (i.e. active) cardiac disease (NYHA Grade II or greater congestive heart failure, symptomatic coronary artery disease, unstable angina, and cardiac arrhythmia not well-controlled with medication), myocardial infarction within the last 6 months prior to study start, or screening ejection fraction of < 50%.
* Any of the following abnormal laboratory values:

  * Absolute neutrophil count < 1.5 x 109/L
  * Platelet count < 100 x 109/L
  * Serum bilirubin > 1.5 x upper limit of normal (ULN)
  * Serum alanine transaminase (ALT), aspartate transaminase (AST) > 2.5 x ULN
  * Serum creatinine > 2.0 mg/dL or 177mmol/L or calculated creatinine clearance by the method of Cockcroft and Gault < 50mL/min).
* Any severe or poorly controlled systemic disease (e.g., hypertension; clinically significant cardiovascular, pulmonary, or metabolic disease, disorders of wound-healing, ulcer or bone fracture).
* Patients who have received any investigational treatment within 4 weeks of study start.
* Known infection with HIV, Hepatitis B virus (HBV), or Hepatitis C virus (HCV).
* Known hypersensitivity to any of the components of NOV-002 or to any of the study drugs.
* Patients assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol.

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-06-04 (Actual); Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keisuke Shirai, MD, Study Chair — Medical University of South Carolina; Alberto Montero, MD, Principal Investigator — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- [Result] Montero AJ, Diaz-Montero CM, Deutsch YE, Hurley J, Koniaris LG, Rumboldt T, Yasir S, Jorda M, Garret-Mayer E, Avisar E, Slingerland J, Silva O, Welsh C, Schuhwerk K, Seo P, Pegram MD, Gluck S. Phase 2 study of neoadjuvant treatment with NOV-002 in combination with doxorubicin and cyclophosphamide followed by docetaxel in patients with HER-2 negative clinical stage II-IIIc breast cancer. Breast Cancer Res Treat. 2012 Feb;132(1):215-23. doi: 10.1007/s10549-011-1889-0. Epub 2011 Dec 3. PMID 22138748

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NOV-002 and Chemotherapy
Started | 41
Completed | 39
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | NOV-002 and Chemotherapy
Number analyzed (Participants) | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 31
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 13
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Rate of Pathologic Complete Response in the Affected Breast After Protocol Therapy
Description: The primary objective of this study is to define the rate of pathologic complete response rate (pCR) in the affected breast after the preoperative administration of NOV-002 in combination with doxorubicin and cyclophosphamide followed by docetaxel in patients with stage IIB-IIIC breast cancer. Pathologic complete response (pCR) is defined according to Hankoop et al [41] as either: the absence of any histological evidence of invasive breast cancer cells in the tissue specimen removed from the breast or the presence of invasive tumor equal to or less than 10mm after preoperative treatment, determined at definitive breast surgery.
Time Frame: About 7 months
Population: Assessable tumors from study participants who had received at least one cycle of protocol therapy.
Measure: Median (95% Confidence Interval); unit: percentage of tumors
Units Other Than Participants: Tumors
Arm/Group | NOV-002 and Chemotherapy
Number analyzed (Participants) | 39
Number analyzed (Tumors) | 40
percentage of tumors | 39 [25 to 45]

2. Secondary Outcome: Definition of the Safety Profiles of Protocol Therapy
Description: Definition of the safety profiles of protocol therapy in study participants as shown by the number of study participants experiencing adverse events or other toxicity.
Time Frame: Up to 30 days Post-Last Dose of Protocol Therapy, About 7 months
Measure: Number; unit: participants
Groups:
- NOV-002 and Chemotherapy: * NOV-002:
    * Cycle 1, Day -1 only: 60 mg intravenously (IV) x 2, 3 hours (+/- 30 minutes) apart
    * Cycles 1 - 8, Day 1: 60 mg IV, 1 hour (+/- 30 minutes) prior to chemotherapy administration
    * Cycle 1 - 8, Days 2 - 21: 60 mg subcutaneous injections
  * Cyclophosphamide: 600 mg/m2 IV, Cycles 1 - 4, Day 1
  * Doxorubicin: 60 mg/m2 IV, Cycles 1 - 4, Day 1
  * Docetaxel: 100 mg/m2 IV, Cycles 5 - 8, Day 1
  Cyclophosphamide
  Docetaxel
  Doxorubicin
  NOV 002
Arm/Group | NOV-002 and Chemotherapy
Number analyzed (Participants) | 41
participants | 41

3. Secondary Outcome: Correlation Between Myeloid Derived Suppressor Cell (MDSC) Levels and Pathologic Complete Response (pCR) and Non-Responders
Description: The investigators hypothesized that patients with favorable responses, i.e. pCR, are more likely to have significantly lower levels of MDSCs than non-responders. MDSC levels will be measured at baseline and on day 1 of each treatment cycle, cycles 1 through 8.
Time Frame: Baseline, Day 1 of Cycles 1 through 8, about 7 months
Population: Study participants who were evaluable for pathologic response.
Measure: Mean (Standard Error); unit: MDSC/uL
Arm/Group | NOV-002 and Chemotherapy
Number analyzed (Participants) | 39
MDSC/uL
  Baseline, non-pCR | 257.4 (0.001)
  Baseline, pCR | 124.3 (0.001)
  Cycles 2-4 Day 1, non-pCR | 534.2 (0.02)
  Cycles 2-4 Day 1, pCR | 207.8 (0.02)
  Cycles 5-8 Day 1, non-pCR | 363.7 (0.006)
  Cycles 5-8 Day 1, pCR | 171.5 (0.006)

ADVERSE EVENTS:
Arm/Group | NOV-002 and Chemotherapy
Serious Adverse Events (participants affected / at risk) | 27/41
Other Adverse Events (participants affected / at risk) | 41/41
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NOV-002 and Chemotherapy (N=41)
Febrile Neutropenia (Blood and lymphatic system disorders) | 4
Sensory Neuropathy (Nervous system disorders) | 4
Abdominal Pain (Gastrointestinal disorders) | 2
Fatigue (General disorders) | 2
Headache (General disorders) | 1
Cellulitis (Musculoskeletal and connective tissue disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1
Deep Vein Thrombosis (Blood and lymphatic system disorders) | 1
Femoral Artery occlusion (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Palmar-plantar erythroysaesthesia (Musculoskeletal and connective tissue disorders) | 6
Pulmonary embolism (Blood and lymphatic system disorders) | 1
Nausea (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NOV-002 and Chemotherapy (N=41)
Nausea (General disorders) | 31
Fatigue (General disorders) | 29
Consitpation (Gastrointestinal disorders) | 16
Vomiting (Gastrointestinal disorders) | 15
Sensory Neuropathy (Nervous system disorders) | 11
Diarrhea (Gastrointestinal disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes